CLINICAL TRIAL: NCT05333042
Title: External Validation of a Deep Learning Based Model for Pulmonary Embolism Detection on Chest CT Scans
Status: Completed | Type: Observational
Sponsor: OncoRadiomics (Industry)
Collaborators: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Sponsor
Other Study IDs: 0156_PE detector validation
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-04

CONDITIONS: Pulmonary Embolism
Keywords: AI, Deep learning, Pulmonary embolism, CT scan
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The scope of this study is the external validation of an explainable deep learning-based classifier for the diagnosis and detection of pulmonary embolism in computed tomography pulmonary angiography (CTPA) and contrast enhanced CT scans.

DETAILED DESCRIPTION:
Pulmonary embolism (PE) is a potentially fatal disease if not promptly diagnosed and treated. Chest CTPA remains the gold standard for diagnosis nowadays, but PE can also be incidentally found on enhanced CT scans. Most CTPA exams are performed in clinics in case of suspicion of PE in urgent conditions, whereas a minority is performed for conditions of suspicious or validated chronic pulmonary thromboembolism, a disease frequently overlooked on CT scans but affected by high morbidity and poor prognosis if left untreated. Thus methods to expedite and automatize the recognition of emboli within pulmonary vessels have the potential of becoming an important support in clinical practice, enabling the better triage of urgent cases of PE and an increased sensitivity in the identification of patients with chronic pulmonary thromboembolism. Based on these clinical needs, a deep learning-based model for the detection of pulmonary embolism has been developed on CTPA scans. The model was based on 2D ResNext50 architecture and was trained and validated using a multicentric open source dataset composed of 7169 patients. From these retrospective data, 85,000 slices positive for PE and 123,428 negative for PE were extracted for training. For internal validation, 9,922 slices were used for each class. The model was initially externally validated at the patient-level using a dataset of 156 adult patients from 3 different public sources, with all emboli segmented by at least one experienced radiologist. To gain insight into the model predictions, activation maps were extracted using the Grad-CAM method. Comparing these maps with the ground truth (GT) segmentations, it was determined if the activated regions corresponded to regions of PE by computing the percentage of GT PE that was activated and the percentage of activated regions corresponding to GT PE. The PE classification model reached an area under the curve (AUC) of 0.86 [0.800-0.919], a sensitivity of 82.68 % [75.16 - 88.27] and a specificity of 79.31 % [61.61 - 90.15] on the external validation set. However, these results have been obtained in an unbalanced external validation cohort (127 PE positive against 29 PE negative patients), thus it is very important to assess the model performances also in a more balanced patients cohort, representing the real clinical incidence of PE (between 12 and 22%). For this reason the scope of the present study is to collect an external validation cohort representative of the real clinical reality, including both CTPA and enhanced CT scans, with a more balanced percentage of positive and negative PE cases. Moreover, the performances of the model will be compared between enhanced CT and CTPA scans.

ELIGIBILITY:
Inclusion Criteria:

* Any patient that has benefit from contrast enhanced CT scan for any clinical reason
* Availability of contrast enhanced images with standard reconstruction kernel and at mediastinal window

Exclusion Criteria:

* Opposition to participate to retrospective clinical trial
* Severe respiratory and hard beam artifacts
* Patients already included in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is composed of participants who underwent an enhanced chest CT scan for screening purposes for the suspicion of pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
The detection performances of the deep learning model | baseline
  Area under the curve (AUC), sensitivity and specificity for the deep learning model in the identification of pulmonary embolism on enhanced chest CT scan

SECONDARY OUTCOMES:
Comparison of performances of the deep learning model on CTPA and enhanced CT scans | baseline
  Area under the curve (AUC), sensitivity and specificity for the deep learning model in the identification of pulmonary embolism on enhanced chest CT scan compared to the CTPA scans

CONTACTS AND LOCATIONS:
Overall Officials: Paul Meunier, PhD, Principal Investigator — CHU of Liege
Locations (1):
- Hospital Center Universitaire De Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No